CLINICAL TRIAL: NCT06267846
Title: A Phase 2, Multicenter, Randomized, Double-Blind, Placebo-Controlled Study to Assess the Efficacy, Safety, and Tolerability of NBI-1070770 in Adults With Major Depressive Disorder
Brief Title: A Study to Evaluate the Efficacy and Safety of NBI-1070770 in Adults With Major Depressive Disorder
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Neurocrine Biosciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: NBI-1070770-MDD2029
Record Dates: First submitted 2024-02-12; First posted 2024-02-20 (Actual); Last update posted 2025-10-29 (Actual); Status verified 2025-10

CONDITIONS: Major Depressive Disorder
Keywords: Major Depressive Disorder; MDD; NBI-1070770; Neurocrine; Antidepressant; Depression; Montgomery-Åsberg Depression Rating Scale; MADRS
MeSH Terms: conditions — Depressive Disorder, Major; Depression

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- NBI-1070770: Low Dose (Experimental): Participants will receive low-dose NBI-1070770.
  Interventions: Drug: NBI-1070770
- NBI-1070770: Medium Dose (Experimental): Participants will receive medium-dose NBI-1070770.
  Interventions: Drug: NBI-1070770
- NBI-1070770: High Dose (Experimental): Participants will receive high-dose NBI-1070770.
  Interventions: Drug: NBI-1070770
- Placebo (Placebo Comparator): Participants will receive matching placebo.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: NBI-1070770 — Suspension for oral administration
  Arms: NBI-1070770: High Dose; NBI-1070770: Low Dose; NBI-1070770: Medium Dose
Drug: Placebo — Suspension for oral administration
  Arms: Placebo

SUMMARY:
To evaluate the efficacy, safety, and tolerability of NBI-1070770 compared to placebo on improving symptoms of depression in participants with major depressive disorder (MDD).

ELIGIBILITY:
Key Inclusion Criteria:

Participants must meet all of the following inclusion criteria:

* Primary diagnosis of recurrent MDD or persistent MDD.
* Participants currently receiving pharmacological treatment for depression must have been taking current antidepressant medication(s) for ≥8 weeks prior to screening and must be willing and able to continue with current antidepressant medication(s).
* Participants must be willing and able to comply with all study procedures and restrictions.

Key Exclusion Criteria:

Participants will be excluded from the study if they meet any of the following criteria:

* Participant is pregnant or breastfeeding or plan to become pregnant during the study.
* Participant has an unstable medical condition or unstable chronic disease.
* Participant has a history of neurological abnormalities.
* Participant has a current or prior psychiatric disorder diagnosis that was the primary focus of treatment other than MDD.
* Participant's depressive symptoms have previously demonstrated nonresponse to an adequate course of treatment with electroconvulsive therapy.
* Participant has an alcohol or substance use disorder.

Note: Other inclusion/exclusion criteria may apply

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 73 (Actual)
Dates: Start 2024-03-20 (Actual); Primary Completion 2025-07-25 (Actual); Study Completion 2025-09-11 (Actual)

PRIMARY OUTCOMES:
Change in Total Montgomery-Åsberg Depression Rating Scale (MADRS) Score from Baseline to Day 5 | Baseline, Day 5

SECONDARY OUTCOMES:
Change in Total MADRS Score from Baseline at Postbaseline Timepoints | Baseline, up to Day 49

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Development Lead, Study Director — Neurocrine Biosciences
Locations (13):
- United States (13):
  - Neurocrine Clinical Site, Little Rock, Arkansas
  - Neurocrine Clinical Site, Rogers, Arkansas
  - Neurocrine Clinical Site, Lemon Grove, California
  - Neurocrine Clinical Site, Long Beach, California
  - Neurocrine Clinical Site, Hollywood, Florida
  - Neurocrine Clinical Site, Maitland, Florida
  - Neurocrine Clinical Site, Decatur, Georgia
  - Neurocrine Clinical Site, Savannah, Georgia
  - Neurocrine Clinical Site, Gaithersburg, Maryland
  - Neurocrine Clinical Site, Dayton, Ohio
  - Neurocrine Clinical Site, North Canton, Ohio
  - Neurocrine Clinical Site, Houston, Texas
  - Neurocrine Clinical Site, Richardson, Texas

IPD SHARING:
Plan to Share IPD: No